CLINICAL TRIAL: NCT03378154
Title: Intubation Success and Glottis Visualization With King Vision Video Laryngoscope as Compared to Conventional Laryngoscopes in Children < 1 Years: A Randomized Control Trial
Brief Title: Comparing the Efficacy of King Vision in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jawaharlal Institute of Postgraduate Medical Education & Research (Other Government)
Responsible Party: Principal Investigator, M Manov, Principal investigator, Jawaharlal Institute of Postgraduate Medical Education & Research
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JIP/IEC/2017/0273
Record Dates: First submitted 2017-11-08; First posted 2017-12-19 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Orotracheal Intubation in Infants Requiring General Anaesthesia for Surgery
Keywords: King vision; Difficult airway; Videolaryngoscope; Paediatric intubation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tracheal Intubation in infants using Macintosh laryngoscopes (Experimental): Children < 1 year of age posted for elective or emergency surgical procedure will be administered general anaesthesia by means of orotracheal intubation with the help of the Macintosh laryngoscope
  Interventions: Procedure: Orotracheal intubation in infants with Macintosh
- Tracheal Intubation in infants using King vision (Experimental): Children < 1 year of age posted for elective or emergency surgical procedure will be administered general anaesthesia by means of orotracheal intubation with the help of the King vision videolaryngoscope
  Interventions: Procedure: Orotracheal intubation in infants with King vision

INTERVENTIONS:
Procedure: Orotracheal intubation in infants with Macintosh — Orotracheal intubation in infants using Macintosh laryngoscope
  Arms: Tracheal Intubation in infants using Macintosh laryngoscopes
Procedure: Orotracheal intubation in infants with King vision — Orotracheal intubation in infants with King vision videolaryngoscope
  Arms: Tracheal Intubation in infants using King vision

SUMMARY:
The primary objective of this study is to find out whether the intubation success rates of Kingvision video laryngoscope is better than that of the conventional laryngoscopes in children < 1 year of age?

DETAILED DESCRIPTION:
Securing the airway by tracheal intubation is one of the most critical steps during administration of general anesthesia to infants. Failure or a delay in tracheal intubation leads to severe hypoxic insult to infants as the oxygen consumption is high in them when compared to adults.Smaller caliber of the pediatric airway, relatively large tongue, anteriorly located larynx, floppy and relatively large epiglottis predispose young children to airway obstruction during Anaesthesia. In addition, the large occiput of the infant places the head and neck in the flexed position when the patient is placed recumbent, further exacerbating airway obstruction

Direct laryngoscopy requires a direct line of sight for proper glottis visualization which is achieved by proper alignment of airway axes (oral-pharyngeal-laryngeal). These manipulations can lead to significant hemodynamic disturbance, cervical instability, injury to oral and pharyngeal tissues and dental damage. In contrast to direct laryngoscopy, video laryngoscope utilizes indirect laryngoscopy via its camera and helps improve glottic visualization, thereby minimizing complications

New age videolaryngoscopes with their unique design provide better glottis visualization without the requirement of proper alignment of oral-pharyngeal-laryngeal axes, thereby minimizing the complications associated with excessive manipulation and hence provide a decent edge over the conventional indirect laryngoscopes routinely used. With the above mentioned advantages these videolaryngoscopes can be efficiently used in both elective as well as emergencysettings in infants for intubation The investigators in this study will be evaluating the efficacy of King vision video laryngoscope when compared to the conventional laryngoscopes in routine use for infants.

ELIGIBILITY:
Inclusion Criteria

* Patients of the age group 0-1 years undergoing elective or emergency surgeries belonging to American Society ofAnaesthesiologists(ASA) physical status classification 1-2 and requiring administration of General Anaesthesia with orotracheal intubation

Exclusion Criteria:

* Patients with anticipated difficult airways
* Patients with aspiration risk or requiring Rapid sequence induction (RSI)
* Patients with laryngeal or tracheal pathologies
* Cervical spine injury
* Active respiratory infection or lung disease

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
First attempt intubation success rate | 0 - 15 minutes
  Comparison of first attempt intubation success rate of King vision videolaryngoscope and the Macintosh laryngoscope in children < 1 year. A total of two laryngoscopy attempts each lasting not more than 60 secs will be allowed. Inability to secure the airway by means of successful orotracheal intubation within the 2 attempts will be taken as a failure. Success rates of both the devices will be compared in the study.

SECONDARY OUTCOMES:
Cormack-Lehane grading (CL grade) | 0 - 15 minutes
  Comparison of Cormack-Lehane grading using King vision and Macintosh laryngoscope. CL grading is a 4 point grading system used to classify the glottic view obtained while performing laryngoscopy (CL 1,2,3,4). A better CL grade obtained is associated with a higher success rate. CL grade obtained with both the devices will be compared in the study.
Percentage of glottic opening score (POGO score) | 0 - 15 minutes
  Comparison of POGO scoring(with and without BURP manuever) using King vision and Macintosh laryngoscope will done in he study
Ease of insertion | 0 - 15 minutes
  Comparison of ease of insertion of King vision and Macintosh laryngoscope will be done based on a 5 point Likert scale.
Mean intubation time | 0 - 15 minutes
  Comparison of Mean intubation time of King vision video laryngoscope and Macintosh laryngoscope in children< 1 year of age. Mean intubation time will be taken as the time between the scope passing the teeth to the appearance of the first end tidal Co2(EtCo2) curve.

CONTACTS AND LOCATIONS:
Locations (1):
- JIPMER, Puducherry, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shravanalakshmi D, Bidkar PU, Narmadalakshmi K, Lata S, Mishra SK, Adinarayanan S. Comparison of intubation success and glottic visualization using King Vision and C-MAC videolaryngoscopes in patients with cervical spine injuries with cervical immobilization: A randomized clinical trial. Surg Neurol Int. 2017 Feb 6;8:19. doi: 10.4103/2152-7806.199560. eCollection 2017. PMID 28217398
- [Background] Sinha R, Sharma A, Ray BR, Kumar Pandey R, Darlong V, Punj J, Chandralekha C, Upadhyay AD. Comparison of the Success of Two Techniques for the Endotracheal Intubation with C-MAC Video Laryngoscope Miller Blade in Children: A Prospective Randomized Study. Anesthesiol Res Pract. 2016;2016:4196813. doi: 10.1155/2016/4196813. Epub 2016 May 15. PMID 27293429
- [Background] Holm-Knudsen RJ, Rasmussen LS. Paediatric airway management: basic aspects. Acta Anaesthesiol Scand. 2009 Jan;53(1):1-9. doi: 10.1111/j.1399-6576.2008.01794.x. PMID 19128325